CLINICAL TRIAL: NCT04983693
Title: Dementia-Friendly Faith Villages to Support African American Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Fayron Epps, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00114202
Record Dates: First submitted 2021-07-22; First posted 2021-07-30 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Dementia
Keywords: Dementia family caregiver
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This study will recruit 45 dyads of African American family caregivers and African American persons living with dementia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia-friendly Worship Service (Experimental): Caregiver and persons living with dementia dyads attending six dementia-friendly worship services in person or online.
  Interventions: Behavioral: Dementia-friendly Worship Service

INTERVENTIONS:
Behavioral: Dementia-friendly Worship Service — Key elements of dementia-friendly worship services include familiar hymns, prayers and bible stories and short sermons. Participants can attend the worship services either in person or through online video streaming. Participant dyads should watch the six worship services together, over a span of 6 to 8 weeks.

SUMMARY:
The purpose of this project is to develop and test the feasibility and preliminary effects of a program to enhance the capacity of predominantly African American churches to support congregants and their family caregivers who are living with dementia. In particular, this project will examine how dementia-friendly faith village worship services support the well-being of caregivers and care recipients in two African American churches.

DETAILED DESCRIPTION:
Historically, churches have been the backbone of support for African American families. As a source of informal support, affiliations with churches serve as an extension to the family, providing social support to older African Americans not always available from close family and friends. African Americans often turn to their church and worship services for support when in distress. In recent years, the question that often arises is: "Are African American faith communities living out components of their church doctrine in relation to their love and commitment to one another?" Surprisingly, many African American churches do not have programs to support their congregation's aging-in-community or the families and congregants living with dementia.

African Americans are more likely than other racial/ethnic groups to be diagnosed with Alzheimer's disease or other forms of dementia, and 20% of persons living with dementia will be African American by 2050. Similarly, the number of their family caregivers will rapidly grow over the next 20 years. Currently, approximately 15 million family caregivers in the United States serve as significant care resources for persons living with dementia. Persons living with dementia experience progressive distress and confusion, which produces emotional strain, burden, social isolation, and depression for caregivers. This underscores the need to strengthen support services and identify resources and meaningful activities that promote physical and mental well-being for African American family caregivers and community-dwelling persons living with dementia.

Dementia restricts the person and the caregiver from participating in religious communities and familiar religious practices; both become increasingly uncomfortable in church settings due to fear of embarrassment, uncertainty about the person's behavior, and even stigma. The caregiving experience often leads to social isolation as caregivers devote all of their time to their family members, thus diminishing their ability to attend church and experience an atmosphere that can support them. Churches can also provide opportunities for individuals living with dementia to continue living in meaningful ways. Along with the setting, socializing with others can be a great strength for these individuals and their family members. Faith-based institutions play a significant role in the lives of individuals living with dementia, primarily through being present for them and the family members to support their quality of life. Research has shown separate benefits for caregivers attending church and the role religion plays in elders living with dementia. However, there is little work exploring how participation in religious practices together (caregiver and person living with dementia) might promote quality of life for these families. A dementia-friendly faith village worship service could provide a culturally organic way for such families to retain connection with a powerful social network.

This study will take place in the south Atlanta Metropolitan area. Two predominantly African American churches from Fulton and Fayette counties have been identified and are eager and enthusiastic to participate in this project. Interested caregivers will be screened for family eligibility via phone. If eligible, times will be scheduled to consent in person prior to data collection. Those consenting will agree to take part in baseline data collection, attend six dementia-friendly worship services in person or online, provide post-intervention data, and take part in more in-depth qualitative interviews. Caregivers will complete surveys and take part in interviews, while only observational data will be collected for persons living with dementia (PLWD).

ELIGIBILITY:
Inclusion Criteria for Caregivers:

* at least 18 years of age
* caring (4 hours/per day of unpaid assistance) for a community-dwelling family or friend experiencing memory impairment
* able to read, speak, and understand English

Inclusion Criteria for Persons Living With Dementia:

* community-dwelling with memory impairment
* have a family caregiver willing to participate

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Zarit Burden Inventory Score | Baseline, Post-intervention (up to 8 weeks)
  The Zarit Burden Interview is a 22-item scale of objective and subjective caregiver burden. Responses are given on a 5-point scale where 0 = never and 4 = nearly always. Total scores range from 0 to 88 where higher scores indicate greater feelings of being burdened with providing care.
Change in Expressive Support Scale Score | Baseline, Post-intervention (up to 8 weeks)
  Socioemotional support is assessed with the Expressive Support Scale. This instrument includes 8 items measuring the amount of help and support that caregivers receive from relatives and friends. Responses are given on a 4-point scale where 1 = strongly disagree and 4 = strongly agree. Total scores range from 8 to 32 and higher scores indicate greater support.
Change in Positive Appraisal of Care Score | Baseline, Post-intervention (up to 8 weeks)
  Consequential gain is assessed with the Positive Appraisal of Care Scale. This instrument includes 6 items asking about personal, positive aspects of being a caregiver. Responses are given on a 4-point scale where 0 = not at all applicable and 3 = very much applicable. Total scores range from 0 to 18, where higher scores indicate greater positive consequential gain from caregiving.
Change in Dyadic Relationship Scale Caregiver Version Score | Baseline, Post-intervention (up to 8 weeks)
  The caregiver version of the Dyadic Relationship Scale includes 11 items which are responded to on a 4-point scale where 1 = strongly disagree and 4 = strongly agree. There are two subscales which assess dyadic strain (5 items) and positive dyadic interaction (6 items). Total scores for the dyadic strain subscale range from 5 to 20 and higher scores indicate greater levels of strain. Total scores for the positive dyadic interaction subscale range from 6 to 24 and higher scores indicate greater positive interactions.
Change in Revised Memory and Behavior Problem Checklist (RMBPC) Frequency Score | Baseline, Post-intervention (up to 8 weeks)
  The RMBPC is a 24-item scale reporting on frequency of disturbing care recipient behaviors and severity or caregiver reactions to these behaviors. Respondents indicate how frequently problems have occurred on a 5-point scale where 0 = never occurred and 4 = daily or more often. Total frequency scores range from 0 to 96 with higher scores indicating greater frequency of memory and behavior problems exhibited by the PLWD.
Change in Revised Memory and Behavior Problem Checklist (RMBPC) Reaction Score | Baseline, Post-intervention (up to 8 weeks)
  The RMBPC is a 24-item scale reporting on frequency of disturbing care recipient behaviors and severity or caregiver reactions to these behaviors. Respondents indicate the degree to which problems have bothered or upset them on a 5-point scale where 0 = not at all and 4 = extremely. Total reaction scores range from 0 to 96 with higher scores indicating more bothered or upset by memory and behavior problems exhibited by the PLWD.
Observation During Worship Service | Up to 8 weeks
  For in person worship services, observations will focus on interactions within the dyads, interactions of caregivers with church leaders and members of the congregation, and interactions of the PLWD with church leaders and the congregation. For online worship services the observations will focus on interactions within the dyads, and the response to the service of the PLWD. Observations of actions during the worship services are assessed qualitatively and a summary score is not determined.

SECONDARY OUTCOMES:
Post-intervention Interview | At the end of the intervention (up to 8 weeks)
  A subsample of 15 to 20 caregivers will be asked to participate in an hour-long, qualitative interview to provide in-depth understanding of the feasibility and efficacy of the intervention. There is not a summary score for the interview questions.

CONTACTS AND LOCATIONS:
Overall Officials: Fayron Epps, PhD, RN, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available for sharing beginning 3 months and ending 5 years following article publication from this study.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims in the approved proposal. Proposals should be directed to fepps@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website.